CLINICAL TRIAL: NCT02058316
Title: Bronchoalveolar Lavage Lateral-Flow Device Test for Invasive Pulmonary Aspergillosis: a Multicenter Study
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Collaborators: Medical University of Vienna (Other); Medical University Innsbruck (Other); Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Robert Krause, MD, Univ. Prof., Medical University of Graz
Other Study IDs: 25-221
Record Dates: First submitted 2014-01-20; First posted 2014-02-10 (Estimated); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Invasive Pulmonary Aspergillosis
MeSH Terms: conditions — Invasive Pulmonary Aspergillosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients at risk for IPA
  Interventions: Device: Lateral Flow Device Test

INTERVENTIONS:
Device: Lateral Flow Device Test — Testing of leftover BAL samples from clinical routine by the lateral flow device test

SUMMARY:
Background Invasive pulmonary aspergillosis (IPA) remains an important cause of morbidity and mortality among patients with hemato-oncological malignancies. Due to the crude mortality of >90% in absence of adequate treatment, timely diagnosis and early start of antifungal therapy are key factors in the successful treatment of IPA. Various studies have shown that early initiation of antifungal therapy may improve IPA survival to above 70%. Diagnosis of IPA, however, remains difficult as clinical signs and symptoms as well as radiological findings are often unspecific and conventional culture methods lack sensitivity. In recent years antigen testing has therefore become one of the cornerstones of IPA diagnostics. Brochoalveolar lavage (BAL) Galactomannan (GM) testing is currently the most promising approach for early detection of pulmonary infections by this fungus. However, limitations of GM detection are assay turn-around time, which varies widely between centers (less than a day to several days), and the need for appropriately equipped laboratories that routinely test for this antigen. These limitations are overcome by the Aspergillus Lateral-Flow Device (LFD), a novel point-of-care (POC) test for IPA diagnosis developed by Dr Thornton at the University of Exeter, UK. This simple, rapid (15 min), single-use test can be performed in rudimentary facilities using BAL specimens. In a retrospective single centre study we have recently evaluated the LFD test in 39 BAL samples from hematologic malignancy patients and solid organ transplant recipients. Sensitivities and specificities of BAL LFD tests for probable IPA were 100% and 81%, respectively. Galactomannan levels in cases with negative LFD were significantly lower than in patients with positive LFD (P <0.0001). We concluded that the LFD test of BAL specimens is performed easily and provides accurate and rapidly available results. Therefore, this new point-of-care test may be a very promising diagnostic approach for detecting IPA in BAL specimens from haematological malignancy and SOT patients. For routine clinical use, however, multicenter studies with larger sample sizes also from other patient collectives are necessary. In this multicenter study we will evaluate the LFD test in BAL samples.

Study Objectives Primary Objectives To evaluate the Lateral Flow Device test, a rapid (15 min), point-of-care test for IPA diagnosis using bronchoalveolar lavage (BAL) fluids from patients at risk for IPA.

Secondary Objective To evaluate the potential of BAL Lateral Flow Device test for prognosis in patients with IPA.

Study Design This is a prospective multi-center study conducted in three centers in Austria (Graz, Vienna and Innsbruck) and one centre in Germany (Mannheim). In order to meet the objectives an estimated number of 300 BAL samples from patients at risk for IPA (50 to 100 per centre) will be included in the study cohort. The Lateral Flow Device test will be performed prospectively in BAL samples from the patients and results will be compared to GM results, PCR findings, clinical/radiological findings as well as conventional culture results. In addition, retrospective testing of BAL samples that were previously routinely tested for GM will be performed in up to three participating centers (Graz, Innsbruck and Mannheim) to ensure to reach the proposed number of 300 BAL samples. The treating clinicians will not be informed about BAL Lateral Flow Device test results and the test will therefore have no impact on patient management / treatment decisions.

DETAILED DESCRIPTION:
Project Outlook Sensitive and specific biomarkers for early diagnosis of IPA are urgently needed to improve survival. In this multicenter study we will evaluate the potential of the novel Lateral Flow Device test for early, bedside diagnosis of IPA.

A successful implementation of the studies hypothesis requires a solid background in the field of IPA. Considering this I am confident that my professional experience combined with the technical and scientific expertise at my host institute and the associated laboratories generates a highly competitive and promising setting. The success of the proposed research will vitally depend on collaborations. Over the last four years I have worked extensively in the field of IPA among patients with hemato-oncological malignancies, which allowed me to establish the necessary contacts and cooperations that are vital for the project's success. The major strength of this multi-center study is therefore the cooperation with three major centers for IPA diagnosis under the leadership of three outstanding experts (Prof. Lass-Flörl, Prof. Buchheidt and Prof. Willinger) who have published extensively in the field of IPA diagnosis over recent years/decades. I am certain that our results will have far-reaching implementations for the whole field of IPA. Clearly, they will significantly advance our understanding of the clinical performance of the novel point of care applications.

The project is expected to have a big impact on patient care. Establishment of the Lateral Flow Device test may lead to rapidly, frankly on the bedside, available test results and may therefore enable earlier initiation of appropriate antifungal therapy which may help to save lives.

1. Background

   Invasive fungal infections (IFI) are an important cause of morbidity and mortality among patients with haemato-oncological malignancies (1-3). Invasive mould infections (IMI), in particular invasive aspergillosis (IA) are the leading cause of IFI among these patients, followed by invasive Candida infections (2, 4). Due to the crude mortality of 80-90% in absence of adequate treatment, timely diagnosis and early start of antifungal therapy are key factors in the successful treatment of IFI. Various studies have shown that early initiation of antifungal therapy may improve IFI survival to above 80% (5, 6). Clinical signs and symptoms of IFI as well as radiological findings, however, are often unspecific. The inability to consistently make an early and convincing diagnosis remains, therefore, one central problem. The European Organization for Research and Treatment of Cancer Invasive Fungal Infections Cooperative Group (EORTC) and the Mycoses Study Group of the National Institute of Allergy and Infectious Disease (MSG) had some success in tackling this problem by establishing consensus definitions for opportunistic IFI (7). However, definitions in EORTC/MSG guidelines were based not only on review of the literature, but also expert opinion and subsequent international consensus. The main reason was that studies evaluating details of the definitions were in part simply not available. In a recent cohort study our working group proposed some modifications to the criteria (8).

   When using EORTC/MSG criteria the prevalence of IFI strongly depends on mycological evidence which is not easy to get. Culture-based diagnostic approaches do not only require invasive diagnostic procedures, which are often hindered by the severe medical condition in patients at risk for IFI, but do also, in fact, frequently result falsely negative. Antigen testing with rapidly available test results has therefore become increasingly important to produce a realistic picture of the burden of IFI and enable early diagnosis and treatment in patients with IFI (1). Antigen testing may not only facilitate early diagnosis but may also prevent overtreatment which has become frequent. A recent study by Azoulay and colleagues who evaluated antifungal therapy on one day in multiple French hospitals confirmed that in fact most of the patients that received antifungals did in fact not have IFI (9). Overtreatment may not only increase costs significantly (daily costs for most antifungals 600-1000€) but may also lead to development of resistance (10). The use of highly sensitive and specific rapidly available antigen tests/ biomarkers may guide the clinician to initiate antifungal therapy only in patients that benefit from treatment as they really have IFI. Last but not least antigen testing may be also useful for early response assessment, therapy monitoring and treatment stratification including the decision when to stop antifungal therapy in patients with IA (11-12).

   One of the major limitations of the GM test is that time to results varies between centres (between less than a day and up to several days), mainly depending on the number of specimens tested in routine (as the test is performed with plates covering 96 tests), and the distance/duration of transport between the clinical setting and the laboratory where the test is performed. These limitations are overcome by the Lateral Flow Device Test, a point of care test for IA developed by Prof. Thornton of the University of Exeter, United Kingdom. This single sample test can be easily performed in every laboratory using BAL and serum specimens and time to result is approximately 20 minutes. Recent studies have shown the immense potential of the test in human BAL and serum samples (13-15). In a very recent study our working group retrospectively evaluated the LFD test by using bronchoalveolar lavage (BAL) samples from patients with haematological malignancies and patients after solid organ transplantation (SOT). Thirty-nine BAL samples from 37 patients were included (29 samples haematological malignancies and 10 samples SOT; 12 probable IPA, 9 possible IPA, 16 no IPA). Sensitivity and specificity of BAL LFD test for probable IPA were 100% and 81%, respectively. GM levels in cases with negative LFD were significantly lower than in patients with positive LFD (P <0.0001). We concluded that the LFD test of BAL specimens is performed easily and provides accurate and rapidly available results. Therefore, this new point-of-care test may be a very promising diagnostic approach for detecting IPA in BAL specimens from haematological malignancy and SOT patients (16). Another recent study demonstrated in a neutropenic guinea pig model that the LFD assay is reproducible between different laboratories and studies (17). Multi-center studies are needed, however, to further evaluate the test (16).

   In the proposed study we will evaluate the BAL Lateral Flow Device Test and compare results to routinely performed Galactomannan values as well as, culture and PCR results.
2. Study design and methods 2.1. Study design The study design is exploratory, retrospective, and multi-centric. The study will start in March 2013 with duration of 13 months.

   2.2. Study sites
   1. Section of Infectious Diseases, Department of Internal Medicine, Medical University of Graz, Austria
   2. Division of Hygiene and Medical Microbiology, Innsbruck Medical University, Austria
   3. Division of Clinical Microbiology, Medical University of Vienna, Austria
   4. Mannheim University Hospital, University of Heidelberg, Germany

   2.3. Study population All stored or routinely obtained BAL samples from adult patients at risk for invasive pulmonary Aspergillosis will be eligible for study inclusion. The treating clinicians will be blinded to BAL Lateral Flow Device test results and the test will therefore have no impact on patient management / treatment decisions. The treating clinicians will be blinded to BAL Lateral Flow Device test results. Test results will therefore have no impact on clinical / treatment decisions and therefore not affect the included patients.

   Underlying diseases, EORTC status of IFI (both available from the clinical order accompanying the BAL sample) and other microbiological/mycological test results will be recorded in an electronic data base. No patient related personal data will be required.

   2.3.1 Key Inclusion criteria
   1. Patients above 18 years of age.
   2. BAL sample obtained in clinical routine.
   3. At risk for IFI (according to attending clinicians). Risk factors may include:

      * febrile neutropenia
      * induction chemotherapy
      * allogeneic stem cell transplant/graft versus host disease
      * clinical/radiological/mycological findings suspicious for IFI
      * Solid Organ transplantation
      * ICU patient
      * Liver cirrhosis 2.3.2 Key exclusion criteria

   <!-- -->

   1. Under 18 years of age.
   2. No BAL sample obtained in clinical routine.

   d.) Not at risk for IFI.

   2.4. Lateral Flow Device testing The previously described lateral flow device is evaluated in BALs from patients at risk for invasive aspergillosis. Briefly, an immunoglobulin G (IgG) monoclonal antibody (JF5) to an epitope on an extracellular antigen secreted constitutively during active growth of Aspergillus is immobilized to a capture zone on a porous nitrocellulose membrane. JF5 IgG is also conjugated to colloidal gold particles to serve as the detection reagent. BAL fluid (100 μl of neat sample, with no pre-treatment) is added to a release pad containing the antibody-gold conjugate, which bound the target antigen, and then passed along the porous membrane and bound to JF5 IgG monoclonal antibody immobilized in the capture zone. Lateral Flow Device (LFD) Results will be read 15 minutes after loading the sample. Bound antigen-antibody-gold complexes are observed as a red line (T for test) with an intensity proportional to the antigen concentration and were classified as negative, weakly positive, moderately positive, or strongly positive (Fig. 1). Anti-mouse immunoglobulin immobilized to the membrane in a separate zone (C for control) serves as an internal control (13, 15). Detailed product information can be found in the attached publication "Development of an Immunochromatographic Lateral-Flow Device for Rapid Serodiagnosis of Invasive Aspergillosis" (14).

   As the device is in the process of being CE marked for European use as a medical diagnostic device, one can only view the current results as a multicentre prototype test comparison (with no clinical implications for patient management).
3. Statistical Considerations Statistical analysis including multivariate analyses will be performed in cooperation with ao. Univ. Prof. Dipl.-Ing. Dr. tech. Josef Haas from the Institute for Medical Informatics, Statistics and Documentation, Medical University of Graz and Univ. Doz. Mag. Dr. Herbert Schwetz, University of Salzburg.

3.1. Sample size calculation Due to the explorative study design statistical sample size calculation is not possible. The samples size has been calculated by using recent published epidemiological data from involved centres (3, 16). The proposed number of patients to be investigated is representative and appropriate to generate data for further studies and has been considered to be adequate by the statistical advisor.

3.2. Statistical Analysis Statistical analysis will be performed by using SPSS in cooperation with our specialized co-operators mentioned above.

References

1. Hoenigl M, Valentin T, Salzer HJ, Zollner-Schwetz I, Krause R. Underestimating the real burden of invasive fungal infections in hematopoietic stem cell transplant recipients? Clin Infect Dis. 2010 Jul 15;51(2):253,4; author reply 254-5.
2. Kontoyiannis DP, Marr KA, Park BJ, Alexander BD, Anaissie EJ, Walsh TJ, et al. Prospective surveillance for invasive fungal infections in hematopoietic stem cell transplant recipients, 2001-2006: Overview of the transplant-associated infection surveillance network (TRANSNET) database. Clin Infect Dis. 2010 Apr 15;50(8):1091-100.
3. Hoenigl M, Salzer HJ, Raggam RB, Valentin T, Rohn A, Woelfler A, et al. Impact of galactomannan testing on the prevalence of invasive aspergillosis in patients with hematological malignancies. Med Mycol. 2012 Apr;50(3):266-9.
4. Perkhofer S, Lass-Florl C, Hell M, Russ G, Krause R, Honigl M, et al. The nationwide austrian aspergillus registry: A prospective data collection on epidemiology, therapy and outcome of invasive mould infections in immunocompromised and/or immunosuppressed patients. Int J Antimicrob Agents. 2010 Dec;36(6):531-6.
5. Greene RE, Schlamm HT, Oestmann JW, Stark P, Durand C, Lortholary O, et al. Imaging findings in acute invasive pulmonary aspergillosis: Clinical significance of the halo sign. Clin Infect Dis. 2007 Feb 1;44(3):373-9.
6. Lass-Florl C, Resch G, Nachbaur D, Mayr A, Gastl G, Auberger J, et al. The value of computed tomography-guided percutaneous lung biopsy for diagnosis of invasive fungal infection in immunocompromised patients. Clin Infect Dis. 2007 Oct 1;45(7):e101-4.
7. De Pauw B, Walsh TJ, Donnelly JP, Stevens DA, Edwards JE, Calandra T, et al. Revised definitions of invasive fungal disease from the european organization for research and treatment of Cancer/Invasive fungal infections cooperative group and the national institute of allergy and infectious diseases mycoses study group (EORTC/MSG) consensus group. Clin Infect Dis. 2008 Jun 15;46(12):1813-21.
8. Hoenigl M, Strenger V, Buzina W, Valentin T, Koidl C, Wolfler A, et al. European organization for the research and treatment of Cancer/Mycoses study group (EORTC/MSG) host factors and invasive fungal infections in patients with haematological malignancies. J Antimicrob Chemother. 2012 May 7.
9. Azoulay E, Dupont H, Tabah A, Lortholary O, Stahl JP, Francais A, et al. Systemic antifungal therapy in critically ill patients without invasive fungal infection*. Crit Care Med. 2012 Mar;40(3):813-22.
10. van der Linden JW, Snelders E, Kampinga GA, Rijnders BJ, Mattsson E, Debets-Ossenkopp YJ, et al. Clinical implications of azole resistance in aspergillus fumigatus, the netherlands, 2007-2009. Emerg Infect Dis. 2011 Oct;17(10):1846-54.
11. Seeber K, Duettmann W, Krause R, Hoenigl M. Usefulness of the serum galactomannan assay for early response assessment and treatment stratifications of invasive aspergillosis. Curr Fungal Infect Rep [DOI: 10.1007/s12281-012-0099-5]. 2012 Online First™, 29 Juni 2012;DOI: 10.1007/s12281-012-0099-5.
12. Chamilos G, Luna M, Lewis RE, Bodey GP, Chemaly R, Tarrand JJ, et al. Invasive fungal infections in patients with hematologic malignancies in a tertiary care cancer center: An autopsy study over a 15-year period (1989-2003). Haematologica. 2006 Jul;91(7):986-9.
13. Thornton C, Johnson G, Agrawal S. Detection of invasive pulmonary aspergillosis in haematological malignancy patients by using lateral-flow technology. J Vis Exp. 2012 Mar 22;(61). pii: 3721. doi(61):10.3791/3721.
14. Thornton CR. Development of an immunochromatographic lateral-flow device for rapid serodiagnosis of invasive aspergillosis. Clin Vaccine Immunol. 2008 Jul;15(7):1095-105.
15. Wiederhold NP, Thornton CR, Najvar LK, Kirkpatrick WR, Bocanegra R, Patterson TF. Comparison of lateral flow technology and galactomannan and (1->3)-beta-D-glucan assays for detection of invasive pulmonary aspergillosis. Clin Vaccine Immunol. 2009 Dec;16(12):1844-6.
16. Hoenigl M, Koidl C, Duettmann W, Seeber K, Wagner J, Buzina W, et al. Bronchoalveolar lavage lateral-flow device test for invasive pulmonary aspergillosis diagnosis in haematological malignancy and solid organ transplant patients. J Infect. 2012;65(6):588-91.
17. Wiederhold NP, Najvar LK, Bocanegra R, Kirkpatrick WR, Patterson TF, Thornton CR. Inter-Laboratory and Inter-Study Reproducibility of a Novel Lateral-Flow Device and the Influence of Antifungal Therapy on the Detection of Invasive Pulmonary Aspergillosis. J Clin Microbiol. 2013; epup ahead of print

ELIGIBILITY:
Inclusion Criteria:

* a.) Patients above 18 years of age. b.) BAL sample obtained in clinical routine. c.) At risk for IFI (according to attending clinicians). Risk factors may include:
* febrile neutropenia
* induction chemotherapy
* allogeneic stem cell transplant/graft versus host disease
* clinical/radiological/mycological findings suspicious for IFI
* Solid Organ transplantation
* ICU patient
* Liver cirrhosis

Exclusion Criteria:

* a.) Under 18 years of age. b.) No BAL sample obtained in clinical routine. d.) Not at risk for IFI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All stored or routinely obtained BAL samples from adult patients at risk for invasive pulmonary Aspergillosis will be eligible for study inclusion. The treating clinicians will be blinded to BAL Lateral Flow Device test results and the test will therefore have no impact on patient management / treatment decisions. The treating clinicians will be blinded to BAL Lateral Flow Device test results. Test results will therefore have no impact on clinical / treatment decisions and therefore not affect the included patients.
  Underlying diseases, EORTC status of IFI (both available from the clinical order accompanying the BAL sample) and other microbiological/mycological test results will be recorded in an electronic data base. No patient related personal data will be required.
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2013-02; Primary Completion 2019-01 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Performance of the Lateral Flow Device Test for diagnosisng of invasive pulmonary aspergillosis in BAL fluids | Day 1
  BAL fluid s of included patients will be tested with the LFD. Results will be compared to other diagnostics.

CONTACTS AND LOCATIONS:
Locations (4):
- Austria (3):
  - Medical university of Graz, Graz
  - Innsbruck medical University, Innsbruck
  - Medical University of Vienna, Vienna
- University Hospital Mannheim, Mannheim, Germany

REFERENCES:
- [Derived] Eigl S, Prattes J, Lackner M, Willinger B, Spiess B, Reinwald M, Selitsch B, Meilinger M, Neumeister P, Reischies F, Wolfler A, Raggam RB, Flick H, Eschertzhuber S, Krause R, Buchheidt D, Thornton CR, Lass-Florl C, Hoenigl M. Multicenter evaluation of a lateral-flow device test for diagnosing invasive pulmonary aspergillosis in ICU patients. Crit Care. 2015 Apr 17;19(1):178. doi: 10.1186/s13054-015-0905-x. PMID 25927915
- [Derived] Prattes J, Flick H, Pruller F, Koidl C, Raggam RB, Palfner M, Eigl S, Buzina W, Zollner-Schwetz I, Thornton CR, Krause R, Hoenigl M. Novel tests for diagnosis of invasive aspergillosis in patients with underlying respiratory diseases. Am J Respir Crit Care Med. 2014 Oct 15;190(8):922-9. doi: 10.1164/rccm.201407-1275OC. PMID 25203869